CLINICAL TRIAL: NCT04164810
Title: Effects of Hydrotherapy on Neuropathic Pain and Pain Catastrophization in Spinal Cord Injury: Study Protocol for a Randomized Controlled Trial
Brief Title: Effects of Hydrotherapy on Neuropathic Pain and Pain Catastrophization in Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad del Valle, Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-1845
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Neuropathic Pain; Spinal Cord Injuries
Keywords: Spinal cord injury; Neuropathic pain; Quality of life; Catastrophization
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Hydrotherapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrotherapy (Experimental): Hydrotherapy intervention will receive the treatment for 9 weeks (2 days per week) , resulting in a total of 18 sessions of Hydrotherapy. Each session will be held for a duration of 45 minutes to 1 hour.
  Interventions: Other: Hydrotherapy
- Physical therapy (Active Comparator): Physical therapy inthervention will have 18 standard physical therapy treatment sessions during 9 weeks. Each session will be held for a duration of 45 minutes to 1 hour.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Hydrotherapy — All sessions will be done by 3 physical therapists specialized in hydrotherapy under different modalities, and a pool equipped to perform this type of intervention. The most commonly used techniques in the institution are Bad Ragaz, for motor control, and the Watsu technique for relaxation and spasticity work.
  Arms: Hydrotherapy
Other: Physical Therapy — All sessions will be done by 3 physical therapists expert in neurorehabilitation, following a physical therapy protocol, which includes stretching, aerobic excercise and muscle strengthening.
  Arms: Physical therapy

SUMMARY:
Spinal Cord Injury (SCI) is a spinal cord injury of traumatic origin with its main etiology being violence, which constitutes one of the greatest social and health problems worldwide. One of the complications with the greatest impact in people with SCI is Neuropathic Pain (NP). Pain, mainly chronic pain, has an effect on emotional states, cognition regarding pain and anticipation which leads to the catastrophization of the pain. This form of pain is related to chronic diseases that develop with pain of poor prognosis and are detrimental to quality of life therefore having enormous impacts on health systems. The physiological mechanisms of Hydrotherapy on pain are clear and there is evidence of its use in the management of painful syndromes of difficult treatments such as that for fibromyalgia and chronic lumbar pain, as well as its positive effect on pain perception. However, the effects of hydrotherapy on the NP of patients with SCI are unknown.

Randomized, controlled clinical trial of parallel groups. A randomized sequence will be carried out in balanced blocks to assign the intervention (Hydrotherapy) or the control (Standard Physical Therapy), to a sample of 28 participants, 14 for each group. Each of the interventions (hydrotherapy and physical therapy) will last 9 weeks, for a total of 18 sessions (2 weekly sessions). Two measurements will be made, baseline (pre-intervention) and a second time one month after the end of the intervention. The validated Spanish scales will be used: NP-4 (NP Screening), Numerical Pain Scale (END), PCS (Pain Catastrophization), SF-36 (Health-related quality of life) and WHODAS 2.0 (Disability). The primary outcome is the level of NP and its catastrophization, and the secondary outcomes are level of disability and quality of life. With 28 participants fully measured, it is possible to have 80% power to find differences between the groups with respect to the primary outcomes. All information will be analyzed using average comparisons with 95% confidence. The analysis will be carried out by Intention to Treat (ITT) taking all the randomized participants. Missing data will be processed through multiple imputation chains. Generalized mixed linear models will be used comparing the standardized baseline and post-intervention averages of each group and between each group, obtaining 95% confidence intervals and p-values. Subgroup analysis will be performed adjusting confounders and interactions. A significant difference will be considered when the value of p is less than 0.05. Cohen´s D will be calculated to identify the size of the intervention effect.

Discussion: The results will reflect the effect of the hydrotherapy on NP in patients with SCI. They will also permit the identification of potential changes in functionality levels or quality of life in the intervened population.

DETAILED DESCRIPTION:
Pain, quality of life and functionality are associated with each other, and patients with SCI are affected by each (4, 5) thus producing limitations in the participation of daily activities and self-care. Pain, mainly chronic pain, has an effect on emotional states as well as cognition regarding pain and anticipation which lead to catastrophization. The previously mentioned is broadly related to chronic diseases that present pain of poor prognosis and are detrimental to quality of life and risk of suicide (6-9) thus having enormous impacts on health systems.

The effects of hydrotherapy in patients with NP secondary to SCI are unknown which is why this study aims to evaluate the effectiveness of hydrotherapy in the decrease of NP, catastrophization of pain, quality of life and disability in a group of patients with SCI.

The main hypothesis of the study is that (i) hydrotherapy is effective in reducing neuropathic pain in patients with NP secondary to SCI. Likewise, another hypothesis to prove is that (ii) hydrotherapy decreases the catastrophization of neuropathic pain in patients with NP secondary to SCI compared to standard physical therapy, and that (iii) hydrotherapy improves the quality of life and the disability of patients with NP secondary to SCI compared to standard physical therapy.

This study is a randomized controlled clinical trial of parallel groups under conditions of usual clinical practice. Participants will be selected from the list of patients attending the Spinal Trauma Clinic of the Physical Medicine and Rehabilitation Unit of a Specialized Trauma Center.

Those eligible for the study are patients whose clinical evaluation and physical examination result in a diagnosis of neuropathic pain secondary to trauma according to the International Spinal Cord Injury Pain (ISCIP), and those that meet the following criteria: over 18 years of age and a DN-score 4 (Douleur Neuropathique-4) equal to or greater than 4 and level of injury below C3.

Those eligible for the study are patients whose clinical evaluation and physical examination result in a diagnosis of neuropathic pain secondary to trauma according to the International Spinal Cord Injury Pain (ISCIP), and those that meet the following criteria: over 18 years of age and a DN-score 4 (Douleur Neuropathique-4) equal to or greater than 4 and level of injury below C3.

Te population requires a medical evaluation, when it is finished, the participants will be randomized into the control and intervention groups. The patient will be informed and reminded via phone call about the first day of therapy initiation.

The comparison groups will be: Intervention Group (Hydrotherapy) and Control Group (Standard Physical Therapy). Participants will be assessed at the following times (Figure 2. Timeline):

1. Measurement 1 - Baseline - At the beginning of the intervention (Both groups start in their respective groups, for 9 weeks).
2. Measurement 2 - At the end of the intervention (one month after the end of the interventions).

The participants assigned to the intervention (hydrotherapy) will receive the treatment for 9 weeks (2 days per week) , resulting in a total of 18 sessions of Hydrotherapy. Each session will be held for a duration of 45 minutes to 1 hour. Likewise, the control group will have 18 standard physical therapy treatment sessions during the same 9 weeks, with the same duration for each session as the hydrotherapy group.

The instruments that will be used are validated worldwide. The DN-4 (Douleur Neuropathique-4 items, to identify the presence of neuropathic pain, scale of catastrophization of pain and intensity of neuropathic pain. Pain Catastrophization Scale (PCS - Pain Catastrophizing Scale) and the Numerical Pain Scale (END) will be used to catastrophization of pain and intensity of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with spinal cord injury.
* Over 18 years of age.
* A DN-score 4 (Douleur Neuropathique-4) equal to or greater than 4.
* level of injury below C3.

Exclusion Criteria:

* Active pressure ulcers
* An E classification in the ASIA (American Spinal Cord Injury Association)
* Cognitive impairment
* Ostomies
* Permanent bladder catheter
* Signs of systemic inflammatory response
* Urinary symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
DN-4 (Douleur Neuropathique-4 items) | it going to be apply in the session number 1 and 18, and the application time is 10 minutes
  consists of 10 items: 7 related to the quality of pain through an interview and the other 3 items through a clinical exam. This questionnaire, which is validated in Spanish (27), consists of descriptions and signs of pain that are evaluated dichotomously (Yes / No) to identify patients who have a high probability of having a neuropathic pain component. The scores of the individual items are added together to obtain a maximum total score of 10, with a cut-off point ≥ 4
Pain Catastrophization Scale (PCS - Pain Catastrophizing Scale) | it going to be apply in the session number 1 and 18, and the application time is 20 minutes
  The PCS is an instrument validated in Spanish for pathologies such as fibromyalgia and amputee patients, which inquires about the thoughts and feelings that arise in the presence of physical pain caused by diseases, wounds, surgeries, etc. This scale has 13 items rated on a Likert scale from 0 to 4 (0 = Nothing at all; 1 = A little; 2 = Moderately; 3 = A lot; 4 = All time)
Numerical Pain Scale (END) | it going to be apply in the session number 1 and 18, and the application time is 1 minute
  used in various clinical settings for multiple health conditions, and measures pain intensity subjectively through a rating of 0 to 10, where 0 means no pain and 10 the worst pain experienced .

SECONDARY OUTCOMES:
Spanish version of the Quality Short-Form Health Survey 36 (SF-36) | it going to be apply in the session number 1 and 18, and the application time is 20 minutes
  It is made up of 36 items distributed in sub-scales of physical functioning, physical role, body pain, general health, vitality, social function, emotional role and mental health, all with Likert questions and dichotomous (Yes / No) questions with the minimum score being 0 and the maximum 100
WHODAS 2.0 questionnaire of the World Health Organization (WHO) | it going to be apply in the session number 1 and 18, and the application time is 10 minutes
  it is used worldwide and inquires about the difficulties that the individual has due to a particular health condition. For this study, the 12-item version will be used, which is made up of a Likert scale ranging from 'no difficulty" (1) to 'extreme difficulty' / 'cannot do it' (5). The scores will be averaged for analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario del Valle "Evaristo García" ESE, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Derived] Campo AR, Pacichana-Quinayaz SG, Bonilla-Escobar FJ, Leiva-Pemberthy LM, Tovar-Sanchez MA, Hernandez-Orobio OM, Arango-Hoyos GP, Mujanovic A. Effectiveness of Hydrotherapy on Neuropathic Pain and Pain Catastrophization in Patients With Spinal Cord Injury: Protocol for a Pilot Trial Study. JMIR Res Protoc. 2022 Apr 29;11(4):e37255. doi: 10.2196/37255. PMID 35486436